CLINICAL TRIAL: NCT01591850
Title: A Randomized, Single-center, Open-label, One-sequence, Two-period Crossover Study in 3 Parts to Investigate the Effects of Multiple Doses of Ketoconazole (Part 1), Rifampicin (Part 2), and Ritonavir-boosted Atazanavir (Part 3) on the PK of a Single Dose of RO5093151 in Healthy Female & Male Subjects
Brief Title: A Drug-Drug Interaction Study of Ketoconazole, Rifampicin and Ritonavir-Boosted Atazanavir With Single-Dose RO5093151 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None
Other Study IDs: BP27852
Record Dates: First submitted 2012-05-03; First posted 2012-05-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Atazanavir Sulfate; Ketoconazole; Rifampin; Ritonavir

ARMS (3):
- 1 Ketoconazole DDI (Experimental)
  Interventions: Drug: RO5093151; Drug: ketoconazole
- 2 Rifampicin DDI (Experimental)
  Interventions: Drug: RO5093151; Drug: rifampicin
- 3 ATZ/r DDI (Experimental)
  Interventions: Drug: RO5093151; Drug: atazanavir; Drug: ritonavir

INTERVENTIONS:
Drug: RO5093151 — Single oral dose
Drug: atazanavir — Multiple oral doses
  Arms: 3 ATZ/r DDI
Drug: ketoconazole — Multiple oral doses
  Arms: 1 Ketoconazole DDI
Drug: rifampicin — Multiple oral doses
  Arms: 2 Rifampicin DDI
Drug: ritonavir — Multiple oral doses
  Arms: 3 ATZ/r DDI

SUMMARY:
This randomized, single-center, open-label, one-sequence, two-period crossover study in three parts will assess the effects of multiple doses of ketoconazole, rifampicin and ritonavir-boosted atazanavir on the pharmacokinetics of a single dose of RO5093151 in healthy male and female volunteers. In Period 1, subjects will receive a single oral dose of RO5093151. In Period 2, subjects will receive a single oral dose of RO5093151 and multiple oral doses of either ketoconazole, rifampicin or ritonavir-boosted atazanavir. Anticipated time on study is up to 8.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 65 years of age. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and complete physical examination
* Body mass index (BMI) 18 to 30 kg/m2
* Females of child-bearing potential must agree to use two effective methods of contraception, including a barrier method and an intrauterine non-hormonal device (set in place at least 3 months before first dosing) for the duration of the study and at least 1 month after last dosing
* Non-smoker for at least 90 days prior to screening

Exclusion Criteria:

* Pregnant or lactating females
* History of drug abuse in the past 2 years, or suspicion of regular consumption of drugs of abuse, or positive result on drugs of abuse test
* History of alcoholism in the past 2 years, or positive alcohol test
* Positive for hepatitis B, hepatitis C or HIV infection
* Systemic , topical, intranasal or inhaled corticosteroid therapy for more than 2 weeks within 3 months prior to screening
* Participation in an investigational drug or device study within 90 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Part 1: Effect of multiple doses of ketoconazole on single-dose pharmacokinetics of RO5093151 and metabolites: Area under the concentration-time curve (AUC) | Pre-dose and up to 72 hours post-dose
Part 2: Effect of multiple doses of rifampicin on single-dose pharmacokinetics of RO5093151 and metabolites: Area under the concentration-time curve (AUC) | Pre-dose and up to 72 hours post-dose
Part 3: Effect of multiple doses of ritonavir-boosted atazanavir on single-dose pharmacokinetics of RO5093151 and metabolites: Area under the concentration-time curve (AUC) | Pre-dose and up to 72 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 6 month
RO5093151 metabolites: Plasma/urine concentrations | Pre-dose and up to 72 hours post-dose
Pharmacodynamics: Area under the effect curve (AUEC) for plasma cortisol/cortisone (Part 1 only) | Pre-dose and up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Merritt Island, Florida, United States